CLINICAL TRIAL: NCT01074892
Title: A Multicenter Study Comparing Mirena and Systemic Progestin for Endometrial Hyperplasia
Brief Title: A Study Comparing Mirena and Systemic Progestin for Endometrial Hyperplasia
Acronym: Mirena
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Helse Nord (Industry); Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK nr 25/2004
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2012-05

CONDITIONS: Endometrial Hyperplasia
Keywords: endometrial hyperplasia treatment MPA per os LNG-IUD
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Medroxyprogesterone Acetate; Medroxyprogesterone; Progestins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MPA 10 mg per oral cyclic for 6 months (Active Comparator): The peroral treatment is used 10 days each month
  Interventions: Drug: Provera (medroxyprogesterone/progestin)
- MPA 10 mg per os continuous 6 months (Active Comparator): Per oral MPA 10 mg is taken daily for 6 months
  Interventions: Drug: Provera (medroxyprogesterone)
- LNG-IUD for 6 months (Active Comparator): Levonorgestrel impregnated IUD is inserted into the uterine cavity and kept in situ for 6 months
  Interventions: Device: Mirena (levonorgestrel)

INTERVENTIONS:
Drug: Provera (medroxyprogesterone/progestin) — 10 mg tablet, 1 tablet per day taken 10 days per month Duration is 6 months
  Other Names: Provera
  Arms: MPA 10 mg per oral cyclic for 6 months
Drug: Provera (medroxyprogesterone) — 10 mg per oral tablet. One tablet per day for 6 months
  Other Names: Provera
  Arms: MPA 10 mg per os continuous 6 months
Device: Mirena (levonorgestrel) — Inserted in the uterine cavity and kept in situ for 6 months
  Other Names: Mirena
  Arms: LNG-IUD for 6 months

SUMMARY:
Randomized controlled multi-center study with three arms including 200 patients with low risk endometrial hyperplasia. After confirmed diagnosis the patients will receive one of the following treatments:

1. Provera (Medroxyprogesterone (MPA)/progestin) 10 mg per oral treatment for 6 months 10 day each cycle,
2. MPA 10 mg continuously for 6 months,
3. Mirena (Levonorgestrel) impregnated IUD for 6 months.

DETAILED DESCRIPTION:
Background:

Endometrial cancer is the most common gynecologic cancer in the Western world and the incidence is still increasing. Endometrial cancer is principally developing through preliminary stages called endometrial hyperplasia and 10-30 per cent will develop into carcinoma when left untreated. The incidence of endometrial cancer in Norway is presently about 650 cases per year and about 3000 cases of endometrial hyperplasia are estimated. Thus,correct and optimal treatment of endometrial hyperplasia will contribute to prevent endometrial cancer development and also in the long term, to reduce the incidence of endometrial cancer. Correct treatment of endometrial hyperplasia includes operative treatment with hysterectomy of the high risk cases and conservative treatment and follow up for patients with lower risk. As diagnostics of endometrial hyperplasia has been a challenge to pathologists, overtreatment of patients with low risk of cancer development is unfortunately still a problem. In the present study an objective scoring system, D-score, is used to classify the patients into low and high risk hyperplasia. D-score in an objective morphometric analysis and the scoring system has proved reliable to predict the prognosis of each single case as to cancer development or not. By tradition low risk endometrial hyperplasia is treated conservatively with progestin hormones, however, no national routines really exist according to dose, type of progestin, treatment time or distribution route, however, varying doses of per oral treatment is mostly used.

Progestins hormones are known to have a growth regulatory effect on the uterine mucosa. However, treatment success after per oral therapy has shown that up to 50% are non-responders after per oral treatment. On the other hand a few recent studies have reported successful results after using the LNG-IUD as treatment for endometrial hyperplasia with 100 per cent treatment response.

The levonorgestrel impregnated impregnated intrauterine originally constructed for menorrhagia and contraceptive use, is delivering more than hundred times increased concentration of progesterone to the uterine mucosa compared to per oral therapy. Thus , the favourable treatment is attributable to the increased concentration of progestins obtained in the uterine mucosa. Another advantage is that treatment can last for years and that side-effects seen for per oral treatment after progestin therapy can be avoided.

Inclusion:

Most of the patients in the present study are seeing their gynecologist due to irregular bleedings.Biopsy is routinely taken by the gynecologist to exclude malignancy or verify hyperplasia. The biopsy is investigated routinely by a the local pathologist. If the diagnosis of hyperplasia is verified and the patient fulfils the inclusion criteria, the histological specimen is sent to the laboratory in Tromsø for D-score. When D-score is >0, the patient may be included in the study.

D-score:

The D-score system is dividing the patients into three risk groups:

1. Patients having a D-score <0 are shown to have a high risk of cancer development are recommended hysterectomy.
2. Patients having D-score >1 have very low risk of cancer development and are recommended progestin treatment.
3. Patients having D-score 0-1 have an uncertain risk of cancer development and may be treated conservatively. Only patients with D-score > 0 may be included in the study.

Randomization:

When the gynecologist receive the diagnosis and the D-score results and the D-score is in accordance with the inclusion criteria, the patients is asked by her gynecologist to be included in the study.

If consent is given, the randomization is performed by telephone contact with the randomization office , UNN, Tromsø, after written informed consent. The patient is free to leave the study any time without argument.

Treatment:

After randomization the treatment according to assigned treatment arm can be started. During the therapy period the patient will be controlled with repeat biopsy after 3 months and at the end of treatment after 6 months. D-score is repeated if hyperplasia persists. If a negative D-score is performed, the patient will have to leave the study. If D-score is still positive the patient will also leave the study, new therapy is then decided by the local gynecologist.

Control:

All patients will be controlled with repeat biopsy every six month for two years after end of therapy. If recurrence of hyperplasia occurs the patient will leave the study and receive other therapy decided by her own gynecologist after repeated D-score.

Side effects:

All side effects which can be related to treatment during treatment and/or follow-up will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial hyperplasia,
* D-score > 0,
* Age 30-70 years,
* No contra-indications against progestin hormones,
* Written consent,
* Patients who have been treated with transcervical resection need a histologically confirmed diagnosis of hyperplasia taken after the TCR

Exclusion Criteria:

* D-score < 0,
* Age < 30 or > 70,
* Increased sensitivity to progestins,
* Pregnancy,
* Infection or cancer in genitalia or mammary gland,
* Liver disease,
* Serious thrombophlebitis.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2005-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Regression of hyperplasia related to treatment arm after 6 months of therapy | Six months

SECONDARY OUTCOMES:
Recurrence of hyperplasia related to treatment arm during follow-up period | Two years
Side effects during treatment | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Ørbo, MD, PhD, Principal Investigator — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

REFERENCES:
- [Background] Kurman RJ, Kaminski PF, Norris HJ. The behavior of endometrial hyperplasia. A long-term study of "untreated" hyperplasia in 170 patients. Cancer. 1985 Jul 15;56(2):403-12. doi: 10.1002/1097-0142(19850715)56:23.0.co;2-x. PMID 4005805
- [Background] Ferenczy A, Gelfand M. The biologic significance of cytologic atypia in progestogen-treated endometrial hyperplasia. Am J Obstet Gynecol. 1989 Jan;160(1):126-31. doi: 10.1016/0002-9378(89)90103-8. PMID 2912075
- [Background] Orbo A, Baak JP, Kleivan I, Lysne S, Prytz PS, Broeckaert MA, Slappendel A, Tichelaar HJ. Computerised morphometrical analysis in endometrial hyperplasia for the prediction of cancer development. A long-term retrospective study from northern Norway. J Clin Pathol. 2000 Sep;53(9):697-703. doi: 10.1136/jcp.53.9.697. PMID 11041060
- [Background] Vereide AB, Arnes M, Straume B, Maltau JM, Orbo A. Nuclear morphometric changes and therapy monitoring in patients with endometrial hyperplasia: a study comparing effects of intrauterine levonorgestrel and systemic medroxyprogesterone. Gynecol Oncol. 2003 Dec;91(3):526-33. doi: 10.1016/j.ygyno.2003.07.002. PMID 14675671
- [Background] Nilsson CG, Haukkamaa M, Vierola H, Luukkainen T. Tissue concentrations of levonorgestrel in women using a levonorgestrel-releasing IUD. Clin Endocrinol (Oxf). 1982 Dec;17(6):529-36. doi: 10.1111/j.1365-2265.1982.tb01625.x. PMID 6819901
- [Background] Scarselli G, Tantini C, Colafranceschi M, Taddei GL, Bargelli G, Venturini N, Branconi F. Levo-norgestrel-nova-T and precancerous lesions of the endometrium. Eur J Gynaecol Oncol. 1988;9(4):284-6. PMID 3391204
- [Background] Orbo A, Arnes M, Hancke C, Vereide AB, Pettersen I, Larsen K. Treatment results of endometrial hyperplasia after prospective D-score classification: a follow-up study comparing effect of LNG-IUD and oral progestins versus observation only. Gynecol Oncol. 2008 Oct;111(1):68-73. doi: 10.1016/j.ygyno.2008.06.014. Epub 2008 Aug 6. PMID 18684496
- [Background] Baak JP, Nauta JJ, Wisse-Brekelmans EC, Bezemer PD. Architectural and nuclear morphometrical features together are more important prognosticators in endometrial hyperplasias than nuclear morphometrical features alone. J Pathol. 1988 Apr;154(4):335-41. doi: 10.1002/path.1711540409. PMID 3385513
- [Background] Perino A, Quartararo P, Catinella E, Genova G, Cittadini E. Treatment of endometrial hyperplasia with levonorgestrel releasing intrauterine devices. Acta Eur Fertil. 1987 Mar-Apr;18(2):137-40. PMID 3115027
- [Background] Vereide AB, Kaino T, Sager G, Orbo A; Scottish Gynaecological Clinical Trials Group. Bcl-2, BAX, and apoptosis in endometrial hyperplasia after high dose gestagen therapy: a comparison of responses in patients treated with intrauterine levonorgestrel and systemic medroxyprogesterone. Gynecol Oncol. 2005 Jun;97(3):740-50. doi: 10.1016/j.ygyno.2005.02.030. PMID 15885761
- [Background] Vereide AB, Kaino T, Sager G, Arnes M, Orbo A. Effect of levonorgestrel IUD and oral medroxyprogesterone acetate on glandular and stromal progesterone receptors (PRA and PRB), and estrogen receptors (ER-alpha and ER-beta) in human endometrial hyperplasia. Gynecol Oncol. 2006 May;101(2):214-23. doi: 10.1016/j.ygyno.2005.10.030. Epub 2005 Dec 1. PMID 16325240
- [Background] Moe BT, Vereide AB, Orbo A, Jaeger R, Sager G. Levonorgestrel, medroxyprogesterone and progesterone cause a concentration-dependent reduction in endometrial cancer (Ishikawa) cell density, and high concentrations of progesterone and mifepristone act in synergy. Anticancer Res. 2009 Apr;29(4):1047-52. PMID 19414344
- [Derived] Mittermeier T, Farrant C, Wise MR. Levonorgestrel-releasing intrauterine system for endometrial hyperplasia. Cochrane Database Syst Rev. 2020 Sep 6;9(9):CD012658. doi: 10.1002/14651858.CD012658.pub2. PMID 32909630
- [Derived] Orbo A, Vereide A, Arnes M, Pettersen I, Straume B. Levonorgestrel-impregnated intrauterine device as treatment for endometrial hyperplasia: a national multicentre randomised trial. BJOG. 2014 Mar;121(4):477-86. doi: 10.1111/1471-0528.12499. Epub 2013 Nov 28. PMID 24286192